CLINICAL TRIAL: NCT00559351
Title: Possibilities for Improvement of an Outcome of the Treatment in Squamous Cell Carcinoma of the Thoracic Esophagus - a Multicenter Randomized Clinical Phase III Trial.
Brief Title: RCT on the Combined Modality Treatment of Squamous Cell Carcinoma of the Esophagus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficulty in recruitment
Sponsor: Ministry of Scientific Research and Information Technology, Poland (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6P05C01320; PL SCSR 6P05C01320
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-09

CONDITIONS: Esophageal Neoplasms; Squamous Cell Cancer
Keywords: esophagectomy; chemotherapy; chemoradiotherapy; combined modality therapy
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms, Squamous Cell | interventions — Neoadjuvant Therapy; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- S (Active Comparator): esophagectomy
  Interventions: Procedure: transthoracic esophagectomy 2-field extended lymphadenectomy
- CHTS (Experimental): neoadjuvant chemotherapy followed by esophagectomy
  Interventions: Drug: neoadjuvant chemotherapy (cisplatin, 5-fluorouracil)
- CHRTS (Experimental): neoadjuvant chemoradiotherapy followed by esophagectomy
  Interventions: Radiation: neoadjuvant chemoradiotherapy

INTERVENTIONS:
Procedure: transthoracic esophagectomy 2-field extended lymphadenectomy — right thoracotomy, mobilization of the esophagus, mediastinal lymph node dissection, laparotomy, gastric tube formation, abdominal lymph node dissection, anastomosis in the neck
  Arms: S
Drug: neoadjuvant chemotherapy (cisplatin, 5-fluorouracil) — 21-day combination systemic chemotherapy regimen consisted of a continuous infusion of cisplatin (20mg/m2/day) on days 1-5, 17-21 and 5-fluorouracil at 300mg/m2/day on days 1-21 followed by 3-phase transthoracic esophagectomy with 2-field extended lymphadenectomy after 3 week interval
  Arms: CHTS
Radiation: neoadjuvant chemoradiotherapy — 21-day combination systemic chemotherapy regimen consisted of a continuous infusion of cisplatin (20mg/m2/day) on days 1-5, 17-21 and 5-fluorouracil at 300mg/m2/day on days 1-21 with concurrent external beam fractionated irradiation to a total dose of 30Gy (2Gy fractions on days 1-5, 8-12, 15-19) followed by 3-phase transthoracic esophagectomy with 2-field extended lymphadenectomy after 3 week interval
  Arms: CHRTS

SUMMARY:
The purpose of the study was to test a null hypothesis that a combined modality treatment of esophageal cancer with neoadjuvant chemotherapy or chemoradiotherapy is equivalent to surgery alone and what are the benefits from adding irradiation to chemotherapy in neoadjuvant treatment of esophageal cancer.

DETAILED DESCRIPTION:
The choice of the most beneficial method of treatment in esophageal cancer remains controversial and is the subject of vigorous debate. Surgery is still regarded as the principle modality among treatment strategies, with longterm survival achieved mainly in less advanced cases. More advanced cases, diagnosed more frequently, are more problematic in selection of the optimal therapeutic method. One of the options for improving treatment outcome in patients with advanced esophageal cancer is combined modality treatment with chemo- and chemoradiotherapy. Currently available RCTs have tested preoperative chemotherapy or chemoradiotherapy separately in comparison to surgery alone. Moreover, we do not know from these trials what is the added value of irradiation in a combined modality therapy over a preoperative chemotherapy. Another drawback of available RCTs is combining 2 different biological cancer entities: adenocarcinoma and squamous cell carcinoma of the esophagus as well as carcinoma of the esophagus and gastro-esophageal junction. That were the reasons for designing our trial testing 3 principal modes of esophageal cancer therapy: surgery vs. chemotherapy + surgery vs. chemoradiotherapy + surgery on homogenous population of esophageal cancer patients with single pathological type - squamous cell carcinoma affecting thoracic esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Histopathologically proven, clinically stage II-III (cTNM according to AJCC/UICC classification), primary squamous cell carcinoma of the thoracic esophagus
* Patients' age above 18 years
* General condition with Karnofsky performance status of >70
* Circulatory and pulmonary capacity at normal range (FEV1 >60%; FVC >60%, NYHA I-II, cardiac output >40%)
* Normal function of the bone marrow (RBC >3,5 T/l; PLT >100 G/l)
* Normal renal (creatinine <1.5 of the upper limit) and liver (AST or ALT <2,5 of the upper limit or bilirubin <1,5 of the upper limit) function

Exclusion Criteria:

* Metastatic disease
* Synchronous malignancy
* History of other cancer within 5 years prior to esophageal cancer treatment
* History of allergic reaction to cisplatin of 5-fluorouracil
* Systemic infection
* Pregnancy or female patients in childbearing age without proper contraceptives.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2001-12; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
mean, median, 1-year, 3-year, 5-year overall survival | 5 years

SECONDARY OUTCOMES:
toxicity-related morbidity and mortality | 30-day
postoperative morbidity and mortality | 30-day
clinical and pathological response rates | 60-day
curative resection rate | 30-day

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Wallner, MD, PhD, Principal Investigator — 2nd Department of General, Gastrointestinal Surgery & Surgical Oncology of the Digestive Tract, Medical University of Lublin, Poland
Locations (1):
- 2nd Department of General, Gastrointestinal Surgery & Surgical Oncology of the Digestive Tract, Medical University of Lublin, Poland, Lublin, Lublin Voivodeship, Poland